CLINICAL TRIAL: NCT07018856
Title: The CLEAR Vanguard Feasibility Study: Comparative Evaluation of Novice-Performed Lung Ultrasound Versus Chest X-Ray for Pneumothorax Detection Post-Chest Tube Removal in Cardiac Surgery Patients
Brief Title: Feasibility Study of Novice-Performed Lung Ultrasound for Pneumothorax Detection After Cardiac Surgery
Acronym: CLEARVGRD
Status: Recruiting | Type: Observational
Sponsor: Jacobo Moreno Garijo (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Toronto General Hospital (Other); London Health Sciences Centre (Other)
Responsible Party: Sponsor-Investigator, Jacobo Moreno Garijo, Dr. Jacobo Moreno Garijo, MD, MSc, PhD, FASE - Principal Investigator and Cardiac Anesthesiologist, Sunnybrook Health Sciences Centre; Assistant Professor, University of Toronto, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Other Study IDs: 5321; AFP2024-25-SB (Other Grant/Funding Number: Sunnybrook AFP Innovation Fund Grant 2024-25)
Record Dates: First submitted 2025-05-21; First posted 2025-06-13 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Pneumothorax; Cardiac Surgery; Lung Ultrasound; Chest Tube Removal; Postoperative Complications (Cardiopulmonary)
Keywords: Lung Ultrasound; Pneumothorax Detection; Chest Tube Removal; Cardiac Surgery; Point-of-Care Ultrasound; Postoperative Complication; Bedside Ultrasound; Novice Sonographer; Diagnostic Accuracy; Feasibility Study; Critical Care Ultrasound; Trainee-Performed Ultrasound; Chest X-Ray; Medical Education
MeSH Terms: conditions — Pneumothorax; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-Cardiac Surgery Patients Undergoing Chest Tube Removal: This cohort includes adult patients who have undergone cardiac surgery and are scheduled for chest and/or mediastinal chest tube removal in the cardiovascular intensive care unit. Each participant will undergo a lung ultrasound performed by a trained medical trainee and a standard chest X-ray to assess for pneumothorax. No interventions are assigned; this is an observational comparison of two diagnostic modalities.

SUMMARY:
What is the purpose of this study? This study is being done to find out if medical trainees (such as residents and fellows) can learn to use lung ultrasound to detect a collapsed lung (pneumothorax) after heart surgery.

Who is participating in the study? Adults who have recently had heart surgery and are having their chest tubes removed in the intensive care unit may be able to join.

What will happen during the study? After chest tubes are removed, a trained medical trainee will use a small ultrasound device to check the lungs at the bedside. The patient will also have a chest X-ray, which is the usual test. The results from the ultrasound will be compared to the chest X-ray and reviewed by expert doctors.

What is the goal of the study? The goal is to see if it is possible to train medical trainees to use lung ultrasound safely and accurately in real hospital settings. The results will help plan a larger study in the future.

DETAILED DESCRIPTION:
This is a feasibility study to test whether lung ultrasound can be used by medical trainees to detect pneumothorax (collapsed lung) after heart surgery, instead of using a chest X-ray.

Collapsed lungs can happen after chest tubes are removed, which is a common step after heart surgery. While chest X-rays are usually used to check for this, they can sometimes miss cases or take time to complete. Lung ultrasound is a fast, safe, and radiation-free tool that can be done right at the bedside.

In this study, medical trainees-such as anesthesia residents, critical care fellows, or internal medicine residents-will receive focused training on how to use lung ultrasound. After training, they will perform lung ultrasound exams on patients within two hours after chest tube removal. These results will be compared to chest X-rays, and also reviewed by expert doctors who are blinded to the trainee's findings.

The study will take place at three large hospitals in Ontario, Canada. It will include about 120 patients in total. The study team will look at how well trainees follow the protocol, how accurate their ultrasound readings are, and how patients feel about having ultrasound done at the bedside.

This study does not involve any new treatments or medications. The purpose is to see if lung ultrasound can be safely and effectively performed by trainees, and whether a larger study should be done in the future to confirm its benefits.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Undergoing cardiac surgery
* Scheduled for chest and/or mediastinal chest tube removal in the cardiovascular intensive care unit (CVICU)

Exclusion Criteria:

* Severe chronic lung disease that may impair lung ultrasound interpretation, including:
* Subcutaneous emphysema
* COPD or emphysema with FEV₁ < 50% predicted
* Interstitial lung disease with FEV₁ < 75% predicted
* Documented history of pneumothorax prior to chest tube removal requiring intervention
* Mechanical ventilation at the time of eligibility screening
* Inability to undergo lung ultrasound or chest X-ray (e.g., due to hemodynamic instability or positioning limitations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult patients (18 years or older) who have undergone cardiac surgery and are scheduled for chest and/or mediastinal chest tube removal in the cardiovascular intensive care unit (CVICU). Participants will be recruited from three high-volume cardiac centers in Ontario, Canada: Sunnybrook Health Sciences Centre, Toronto General Hospital, and London Health Sciences Centre. Patients must be able to safely undergo both lung ultrasound and chest X-ray after chest tube removal. Individuals with severe lung disease or who are mechanically ventilated at the time of eligibility screening will be excluded.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate Across Sites | Up to 12 months after study start
  Recruitment feasibility will be measured by the number of participants enrolled per site per month. The target is at least 2 patients per site per month across three participating centers. Unit of Measure: Participants per site per month
Protocol Adherence to Lung Ultrasound Procedures | Up to 12 months after study start
  Percentage of enrolled participants with complete protocol adherence, defined as having both lung ultrasound and chest X-ray performed and documented as per protocol, including all required images and forms. Unit of Measure: Percentage.
Participant Attrition Rate | Up to 12 months after study start
  Percentage of enrolled participants who withdraw or are lost to follow-up before completion of study procedures. The study aims to maintain an attrition rate below 10%. Unit of Measure: Percentage.
Inter-Rater Agreement Between Novice and Expert Ultrasound Reviewers | Up to 12 months after study start
  Inter-rater reliability for lung ultrasound interpretation between novice trainees and expert reviewers, measured using kappa statistics. The target agreement is a kappa ≥ 0.8. Unit of Measure: Kappa statistic.

SECONDARY OUTCOMES:
Diagnostic Agreement Between Novice-Performed Lung Ultrasound and Chest X-Ray for Pneumothorax Detection | Up to 2 hours after chest tube removal on Day 0
  This outcome compares the diagnostic accuracy of lung ultrasound performed by trained medical trainees to standard chest X-ray for pneumothorax detection following chest tube removal. Agreement will be assessed using kappa statistics. Expert reviewers will independently evaluate LUS images while radiologists will interpret CXR images, both blinded to each other's findings.
Time to Diagnosis: Lung Ultrasound vs. Chest X-Ray | Up to 2 hours after chest tube removal on Day 0
  Compare the time from chest tube removal to pneumothorax diagnosis using lung ultrasound versus chest X-ray. Time will be measured in minutes from tube removal to the documented result of each imaging modality.
Patient-Reported Experience With Lung Ultrasound | Immediately after lung ultrasound on Day 0
  Assess patient-reported comfort, acceptability, and imaging preference using a short questionnaire with Likert-scale responses following lung ultrasound.
Adverse Events Related to Missed Pneumothorax | From chest tube removal through hospital discharge (up to 14 days, based on the expected max stay)
  Monitor for complications associated with missed or delayed pneumothorax diagnosis, including respiratory failure, chest tube reinsertion, ICU readmission, or in-hospital mortality.

OTHER OUTCOMES:
Diagnostic Sensitivity and Specificity of Lung Ultrasound vs. Chest X-Ray | Within 2 hours of chest tube removal
  Sensitivity and specificity of novice-performed lung ultrasound will be calculated for pneumothorax detection, using expert-reviewed chest X-ray as the clinical standard.
Image Quality Scores of Trainee-Performed Lung Ultrasound | Immediately following each lung ultrasound (same day as chest tube removal)
  Expert reviewers will assess image quality using a 3-point scale (inadequate, adequate, optimal) for each LUS exam performed by trainees. The proportion of adequate or better images will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Jerath, MD, Study Chair — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
At this time, no decision has been made regarding the sharing of individual participant data (IPD). The primary aim of this study is to assess feasibility and diagnostic accuracy in a small, multicenter pilot cohort. If future analysis supports broader data sharing and aligns with institutional ethics and privacy policies, a data-sharing plan may be developed for the larger, definitive trial.

REFERENCES:
- [Background] McAlinden C, Khadka J, Pesudovs K. Statistical methods for conducting agreement (comparison of clinical tests) and precision (repeatability or reproducibility) studies in optometry and ophthalmology. Ophthalmic Physiol Opt. 2011 Jul;31(4):330-8. doi: 10.1111/j.1475-1313.2011.00851.x. Epub 2011 May 26. PMID 21615445
- [Background] Bland JM, Altman DG. Measuring agreement in method comparison studies. Stat Methods Med Res. 1999 Jun;8(2):135-60. doi: 10.1177/096228029900800204. PMID 10501650
- [Background] Dessie AS, Calhoun AW, Kanjanauptom P, Gilbert GE, Ekpenyong A, Lewiss RE, Rabiner JE, Tsze DS, Kessler DO. Development and Validation of a Point-of-Care-Ultrasound Image Quality Assessment Tool: The POCUS IQ Scale. J Ultrasound Med. 2023 Jan;42(1):135-145. doi: 10.1002/jum.16095. Epub 2022 Sep 27. PMID 36165271
- [Background] Lichtenstein D, Meziere G, Biderman P, Gepner A. The "lung point": an ultrasound sign specific to pneumothorax. Intensive Care Med. 2000 Oct;26(10):1434-40. doi: 10.1007/s001340000627. PMID 11126253
- [Background] Lichtenstein D, Meziere G, Biderman P, Gepner A. The comet-tail artifact: an ultrasound sign ruling out pneumothorax. Intensive Care Med. 1999 Apr;25(4):383-8. doi: 10.1007/s001340050862. PMID 10342512
- [Background] Lichtenstein DA, Menu Y. A bedside ultrasound sign ruling out pneumothorax in the critically ill. Lung sliding. Chest. 1995 Nov;108(5):1345-8. doi: 10.1378/chest.108.5.1345. PMID 7587439
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Volpicelli G. Sonographic diagnosis of pneumothorax. Intensive Care Med. 2011 Feb;37(2):224-32. doi: 10.1007/s00134-010-2079-y. Epub 2010 Nov 20. PMID 21103861
- [Background] Unluer EE, Karagoz A, Oyar O, Vandenberk N, Kiyancicek S, Budak F. Lung ultrasound by emergency nursing as an aid for rapid triage of dyspneic patients: a pilot study. Int Emerg Nurs. 2014 Oct;22(4):226-31. doi: 10.1016/j.ienj.2014.03.003. Epub 2014 Apr 2. No abstract available. PMID 24793725
- [Background] Mumoli N, Vitale J, Giorgi-Pierfranceschi M, Cresci A, Cei M, Basile V, Brondi B, Russo E, Giuntini L, Masi L, Cocciolo M, Dentali F. Accuracy of Nurse-Performed Lung Ultrasound in Patients With Acute Dyspnea: A Prospective Observational Study. Medicine (Baltimore). 2016 Mar;95(9):e2925. doi: 10.1097/MD.0000000000002925. PMID 26945396
- [Background] Shostak E, Brylka D, Krepp J, Pua B, Sanders A. Bedside sonography for detection of postprocedure pneumothorax. J Ultrasound Med. 2013 Jun;32(6):1003-9. doi: 10.7863/ultra.32.6.1003. PMID 23716522
- [Background] Raja AS, Jacobus CH. How accurate is ultrasonography for excluding pneumothorax? Ann Emerg Med. 2013 Feb;61(2):207-8. doi: 10.1016/j.annemergmed.2012.07.005. Epub 2012 Jul 27. No abstract available. PMID 22841178
- [Background] Saucier S, Motyka C, Killu K. Ultrasonography versus chest radiography after chest tube removal for the detection of pneumothorax. AACN Adv Crit Care. 2010 Jan-Mar;21(1):34-8. doi: 10.1097/NCI.0b013e3181c8013a. PMID 20118702
- [Background] Tocino IM, Miller MH, Fairfax WR. Distribution of pneumothorax in the supine and semirecumbent critically ill adult. AJR Am J Roentgenol. 1985 May;144(5):901-5. doi: 10.2214/ajr.144.5.901. PMID 3872573
- [Background] Lin EC. Radiation risk from medical imaging. Mayo Clin Proc. 2010 Dec;85(12):1142-6; quiz 1146. doi: 10.4065/mcp.2010.0260. PMID 21123642
- [Background] Omar HR, Mangar D, Khetarpal S, Shapiro DH, Kolla J, Rashad R, Helal E, Camporesi EM. Anteroposterior chest radiograph vs. chest CT scan in early detection of pneumothorax in trauma patients. Int Arch Med. 2011 Sep 27;4(1):30. doi: 10.1186/1755-7682-4-30. PMID 21951659
- [Background] Galbois A, Ait-Oufella H, Baudel JL, Kofman T, Bottero J, Viennot S, Rabate C, Jabbouri S, Bouzeman A, Guidet B, Offenstadt G, Maury E. Pleural ultrasound compared with chest radiographic detection of pneumothorax resolution after drainage. Chest. 2010 Sep;138(3):648-55. doi: 10.1378/chest.09-2224. Epub 2010 Apr 9. PMID 20382717
- [Background] Roberts DJ, Leigh-Smith S, Faris PD, Blackmore C, Ball CG, Robertson HL, Dixon E, James MT, Kirkpatrick AW, Kortbeek JB, Stelfox HT. Clinical Presentation of Patients With Tension Pneumothorax: A Systematic Review. Ann Surg. 2015 Jun;261(6):1068-78. doi: 10.1097/SLA.0000000000001073. PMID 25563887
- [Background] Bell RL, Ovadia P, Abdullah F, Spector S, Rabinovici R. Chest tube removal: end-inspiration or end-expiration? J Trauma. 2001 Apr;50(4):674-7. doi: 10.1097/00005373-200104000-00013. PMID 11303163
- [Background] Goodman MD, Huber NL, Johannigman JA, Pritts TA. Omission of routine chest x-ray after chest tube removal is safe in selected trauma patients. Am J Surg. 2010 Feb;199(2):199-203. doi: 10.1016/j.amjsurg.2009.03.011. PMID 20113700
- [Background] Khan T, Chawla G, Daniel R, Swamy M, Dimitri WR. Is routine chest X-ray following mediastinal drain removal after cardiac surgery useful? Eur J Cardiothorac Surg. 2008 Sep;34(3):542-4. doi: 10.1016/j.ejcts.2008.05.002. Epub 2008 Jun 9. PMID 18539477